CLINICAL TRIAL: NCT07118930
Title: Prospective Double-Blind Controlled Study of Sivelestat Sodium in the Perioperative Management of Off-Pump Coronary Artery Bypass Grafting
Brief Title: Study of Sivelestat Sodium in OPCABG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-K171-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-06

CONDITIONS: Coronary Heart Disease; Coronary Artery Disease; Coronary Arterial Disease (CAD)
Keywords: coronary heart disease; coronary artery bypass grafting; Sivelestat Sodium; prognosis; myocardial injury
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sivelestat Sodium (Experimental): Sivelestat Sodium injection or a placebo 2 h after OPCABG for 72 h
  Interventions: Drug: Sivelestat Sodium injection 2 h after OPCABG for 72 h
- Routine therapy (Placebo Comparator): Saline instead of Sivelestat
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Sivelestat Sodium injection 2 h after OPCABG for 72 h — Sivelestat Sodium injection 2 h after OPCABG for 72 h
  Arms: Sivelestat Sodium
Drug: Saline (0.9% NaCl) — Saline (0.9% NaCl) instead of Sivelestat
  Arms: Routine therapy

SUMMARY:
The goal of this clinical trial is to learn if drug Sivelestat Sodium works to improve the prognosis of off-pump coronary artery bypass grafting (OPCABG) in adults. It will also learn about the safety of drug Sivelestat Sodium. The main questions it aims to answer are:

* Does drug Sivelestat Sodium have a protective effect on myocardial injury after OPCABG?
* Does Sivelestat Sodium exert a protective effect on myocardial inflammatory stress after OPCABG? Researchers will compare drug Sivelestat Sodium to a placebo (a look-alike substance that contains no drug) to see if drug Sivelestat Sodium works to protect myocardium following OPCABG.

Participants will:

* Accept drug Sivelestat Sodium injection or a placebo 2 h after OPCABG for 72 h.
* Undergo a series of blood tests and echocardiography examinations after the OPCABG.

DETAILED DESCRIPTION:
1.1 Main Objective To evaluate the protective effect of sivelestat sodium on myocardial injury after off-pump coronary artery bypass grafting (OPCABG).

Key observation indicators include: 1) Myocardial injury markers: high-sensitivity cardiac troponin T (hs-cTnT), creatine kinase isoenzyme (CK-MB), NT-proBNP; 2) Cardiac function imaging indicators: global longitudinal strain (GLS) by echocardiography, left ventricular ejection fraction (LVEF).

1.2 Secondary Objective To evaluate the protective effect of sivelestat sodium on myocardial inflammatory stress after OPCABG.

Key observation indicators include: 1) Changes in inflammatory factors (IL-6, CRP, PCT) levels; 2) Observation of clinical outcomes (mechanical ventilation time, ICU stay time, 30-day adverse events, etc.).

2.1 Research Content and Design Prospective, double-blind, randomized, placebo-controlled trial. Prospective design: Standardized data collection from patient enrollment to follow-up completion to avoid recall bias and selection bias in retrospective studies.

Double-blind implementation: Both the subjects, the surgical team, and the outcome assessors are blinded to the group information.

Placebo control: Normal saline for flushing is used as the control to ensure that the basic treatments (anticoagulation, analgesia, etc.) in both groups are completely consistent.

2.2 Research Subjects Patients undergoing elective off-pump coronary artery bypass grafting. 2.3 Research Steps After randomization, the experimental group is administered sivelestat sodium (specification: 0.1 g/vial, Shanghai Huirun Pharmaceutical) at a rate of 0.2 mg/kg/h continuously. Administration starts within 2 hours after surgery and continues for 72 hours. The placebo group is given normal saline for flushing instead of sivelestat sodium. Concomitant medications: Routine anticoagulation and analgesia are allowed, but glucocorticoids or other NE inhibitors are prohibited. The following indicators are measured at preoperative, 2 hours postoperative, 24 hours postoperative, 48 hours postoperative, and 72 hours postoperative: IL-6 (ELISA, R&D Systems), CRP (immunoturbidimetry), CK-MB, cTnI (chemiluminescence); echocardiography is used to assess myocardial motion and cardiac function.

2.4 Evaluation Indicators (Safety, Efficacy Evaluation Criteria, it is recommended to use the latest international or domestic common standards) Efficacy: Primary endpoint (cTnI reduction ≥ 20%); secondary endpoint (IL-6 reduction ≥ 20%).

Safety: Adverse events are recorded using CTCAE 5.0 grading, and their correlation with the study drug is analyzed (see Table in Section 8).

2.5 Data Management and Statistical Analysis Plan, Data Confidentiality Plan An independent data safety monitoring committee (DSMB) is established for data management.

Unblinding conditions: Only independent staff can unblind when serious adverse events (SAEs) require emergency treatment.

Statistical processing software: SPSS 26.0, Graphpad Prism 10. Statistical methods: Intention-to-treat (ITT) analysis, ANCOVA to correct for baseline, measurement data are expressed as mean ± standard deviation, independent sample t-test for comparison between groups, and repeated measures ANOVA for dynamic changes.

3. Subject Recruitment 3.1 Inclusion Criteria Age 18-75 years old, undergoing elective OPCABG (≥2 bypass vessels). LVEF ≥ 35%, no severe liver or kidney function abnormalities (ALT/AST ≤ 3 times the upper limit, eGFR ≥ 60 mL/min).

Signed informed consent form. 3.2 Exclusion Criteria Emergency surgery, combined valve surgery or aortic surgery. Use of immunosuppressants or potent anti-inflammatory drugs within 30 days before surgery.

Active infection, autoimmune disease, or allergy history. Preoperative liver or kidney dysfunction; preoperative severe cardiopulmonary dysfunction.

3.3 Withdrawal and Termination Criteria Withdrawal criteria: Conversion to cardiopulmonary bypass during surgery; postoperative need for IABP, ECMO, or other circulatory support; death or reoperation within 24 hours postoperatively.

Termination criteria: Severe adverse events (SAE, such as anaphylactic shock, liver failure); subject requests withdrawal or is lost to follow-up.

3.4 Duration of Participation for Study Participants (Each Participation Time and Total Time) The total duration of the study is 2 years. Each individual participant's participation period is from 2 hours postoperatively to 72 hours postoperatively, after which the study will be automatically terminated.

3.5 Recruitment Process (Including Recruitment Procedures, Start Time, Methods, Expected Number of Recruits, and Compensation?) Recruitment will commence after study approval, with the first batch expected to start in August 2025.

Recruitment methods include:

In-hospital channels: Posters in the cardiology outpatient department; scrolling display of study introduction on electronic screens (with a QR code linking to detailed information); recommendation by attending physicians during preoperative consultations.

Out-of-hospital channels: Referrals from partner community hospitals; recruitment information pushed on the hospital's official WeChat account (with an online pre-screening questionnaire attached).

Expected number of recruits: 62 cases (31 in the Sivelestat group + 31 in the placebo group); screening ratio: 80 cases expected to be screened, with 20% excluded (emergency surgery, infection, refusal to participate, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective OPCABG (≥2 bridged vessels). LVEF≥35%, no severe liver or kidney function abnormalities (ALT/AST≤3 times the upper limit, eGFR≥60 mL/min). Sign the informed consent form.

Exclusion Criteria:

* Emergency operation, combined valve surgery or aortic surgery. Usage of immunosuppressants or potent anti-inflammatory drugs within 30 days before the operation.
* Active infections, autoimmune diseases, and allergy history.
* Preoperative liver and kidney dysfunction
* Severe cardiopulmonary insufficiency before the operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury | Day 3 after OPCABG
  Sivelestat Sodium exerts a protective effect on myocardial injury after OPCABG

SECONDARY OUTCOMES:
Myocardial inflammatory stress | Day 3 after OPCABG
  Sivelestat Sodium exerts a protective effect on myocardial inflammatory stress after OPCABG

CONTACTS AND LOCATIONS:
Overall Officials: Weizhang Xiao, Dr., Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Basic information, type of operation, experimental results
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Sun L, Zhou M, Ji Y, Wang X, Wang X. Off-pump versus on-pump coronary artery bypass grafting for octogenarians: A meta-analysis involving 146 372 patients. Clin Cardiol. 2022 Apr;45(4):331-341. doi: 10.1002/clc.23794. Epub 2022 Mar 10. PMID 35266173
- [Result] Zhou Y, Li X, Chen H, Zhong X, Ren H. Efficacy and safety of sivelestat sodium for the treatment of inflammatory response in acute Stanford type A aortic dissection: a retrospective cohort study. J Thorac Dis. 2022 Oct;14(10):3975-3982. doi: 10.21037/jtd-22-1220. PMID 36389323
- [Result] Fujii M, Bessho R. Neutrophil Elastase Inhibitor Sivelestat Attenuates Myocardial Injury after Cardioplegic Arrest in Rat Hearts. Ann Thorac Cardiovasc Surg. 2020 Oct 21;26(5):263-269. doi: 10.5761/atcs.oa.19-00240. Epub 2019 Dec 9. PMID 31813921
- [Result] Akiyama D, Hara T, Yoshitomi O, Maekawa T, Cho S, Sumikawa K. Postischemic infusion of sivelestat sodium hydrate, a selective neutrophil elastase inhibitor, protects against myocardial stunning in swine. J Anesth. 2010 Aug;24(4):575-81. doi: 10.1007/s00540-010-0948-8. Epub 2010 May 13. PMID 20464430
- [Result] Sun JK, Li JJ, Deng YH, Yin X, Huangfu XT, Ye ZY, Zhou XH, Chen YM, Yuan ST, Wang X. The beneficial effects of neutrophil elastase inhibitor on gastrointestinal dysfunction in sepsis. Clin Transl Sci. 2024 May;17(5):e13829. doi: 10.1111/cts.13829. PMID 38769746
- [Result] Xu J, Zhang C, Wu K, Qian Y, Hu W. A comparative analysis of sivelestat sodium hydrate and ulinastatin combination therapy in the treatment of sepsis with acute respiratory distress syndrome. BMC Pulm Med. 2024 Jun 17;24(1):283. doi: 10.1186/s12890-024-03083-w. PMID 38886709
- [Result] Henriksen PA. The potential of neutrophil elastase inhibitors as anti-inflammatory therapies. Curr Opin Hematol. 2014 Jan;21(1):23-8. doi: 10.1097/MOH.0000000000000001. PMID 24241342
- [Result] Yu X, Kennedy RH, Liu SJ. JAK2/STAT3, not ERK1/2, mediates interleukin-6-induced activation of inducible nitric-oxide synthase and decrease in contractility of adult ventricular myocytes. J Biol Chem. 2003 May 2;278(18):16304-9. doi: 10.1074/jbc.M212321200. Epub 2003 Feb 20. PMID 12595539
- [Result] Li W, Hsiao HM, Higashikubo R, Saunders BT, Bharat A, Goldstein DR, Krupnick AS, Gelman AE, Lavine KJ, Kreisel D. Heart-resident CCR2+ macrophages promote neutrophil extravasation through TLR9/MyD88/CXCL5 signaling. JCI Insight. 2016 Aug 4;1(12):e87315. doi: 10.1172/jci.insight.87315. PMID 27536731
- [Result] Welt FGP, Batchelor W, Spears JR, Penna C, Pagliaro P, Ibanez B, Drakos SG, Dangas G, Kapur NK. Reperfusion Injury in Patients With Acute Myocardial Infarction: JACC Scientific Statement. J Am Coll Cardiol. 2024 Jun 4;83(22):2196-2213. doi: 10.1016/j.jacc.2024.02.056. PMID 38811097